CLINICAL TRIAL: NCT00887523
Title: Randomized Controlled Trial Comparing Prone and Supine Intensity-modulated Radiotherapy (IMRT) After Breast-conserving Surgery in Patients With Large Breast Volume at High Risk for Skin Toxicity and Fibrosis
Brief Title: Trial Comparing Prone and Supine Intensity-modulated Radiotherapy (IMRT) After Breast-conserving Surgery in Patients With Large Breast Volume at High Risk for Skin Toxicity and Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: National Cancer Plan, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009/184
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2015-06

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation; Prone Position; Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): prone intensity-modulated radiotherapy
  Interventions: Behavioral: radiation in prone position
- 2 (Active Comparator): supine intensity-modulated radiotherapy
  Interventions: Behavioral: radiation in supine position

INTERVENTIONS:
Behavioral: radiation in prone position — radiation in prone position
  Arms: 1
Behavioral: radiation in supine position — radiation in supine position
  Arms: 2

SUMMARY:
84 patients with a cup size C or more will be randomized to receive intensity-modulated radiotherapy in supine or prone position.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* multidisciplinary decision of adjuvant whole-breast irradiation (WBI) after lumpectomy for breast cancer
* minimum 18 years
* informed consent obtained, signed and dated before specific protocol procedures

Exclusion Criteria:

* mastectomy
* need for axillary irradiation
* bilateral breast irradiation
* previous irradiation at the same time
* mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study
* patient unlikely to comply with the protocol; i.e. uncooperative attitude, inability to return for follow-up visits, and unlikely to complete the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
acute moist desquamation | weekly during radiotherapy and 1 month after radiotherapy

SECONDARY OUTCOMES:
Acute skin toxicity other than moist desquamation | weekly during radiotherapy and 1 month after radiotherapy
Late skin toxicity | at 6, 12, 18 and 24 months after radiotherapy
skin and lung fibrosis assessed with computed tomography | before radiotherapy and 1 month and 1 year after radiotherapy
Quality of life | at 1 year and 2 years after radiotherpay
dose-volume parameters | of planning
time of treatment delivery | daily during radiotherapy
single nucleotide polymorphisms associated with skin toxicity and breast fibrosis | 1 blood sample before radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Neve, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Derived] Vakaet V, Van Hulle H, Vergotte M, Schoepen M, Deseyne P, Van Greveling A, Post G, Speleers B, Paelinck L, Monten C, De Neve W, Veldeman L. 5-Year Outcomes of a Randomized Trial Comparing Prone and Supine Whole Breast Irradiation in Large-Breasted Women. Int J Radiat Oncol Biol Phys. 2021 Jul 1;110(3):766-771. doi: 10.1016/j.ijrobp.2021.01.026. Epub 2021 Jan 27. PMID 33508375
- See also: website of the University Hospital Ghent — http://www.uzgent.be